CLINICAL TRIAL: NCT01360918
Title: Concomitant Epicardial Pulmonary Vein Isolation in Patients With Atrial Fibrillation Undergoing Elective Cardiac Surgery
Acronym: CONTROL-AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion rate insufficiënt
Sponsor: Medisch Spectrum Twente (Other)
Collaborators: Foundation of Cardiovascular Research and Education Enschede (Other)
Responsible Party: Principal Investigator, B. Oude Velthuis, B. Oude Velthuis MD., Medisch Spectrum Twente
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL35192.044.11
Record Dates: First submitted 2011-05-13; First posted 2011-05-26 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator)
  Interventions: Other: Usual care
- Pulmonary vein isolation (Active Comparator)
  Interventions: Device: Epicardial pulmonary vein isolation

INTERVENTIONS:
Device: Epicardial pulmonary vein isolation — After the CABG procedure, a bilateral epicardial pulmonary vein isolation is performed under general anaesthesia and double-lumen endotracheal ventilation.
  Other Names: Medtronic Cardioblate BP2
  Arms: Pulmonary vein isolation
Other: Usual care — Management of atrial fibrillation according to current guidelines using rate control pharmacological therapy.
  Arms: Usual care

SUMMARY:
Recent studies demonstrated that radiofrequency isolation of the pulmonary veins (PVI) is a superior alternative to antiarrhythmic drug therapy in patients with symptomatical paroxysmal atrial fibrillation (AF). A substantial proportion of patients undergoing elective cardiac surgery also suffer from atrial fibrillation. No evidence exists if epicardial PVI is beneficial in patients with a history of AF undergoing coronary bypass surgery (CABG) for the concomitant treatment of AF. The investigators aim to establish the effectiveness of incorporating epicardial pulmonary vein isolation into elective cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* EHRA class ≤ 2
* Documented history of paroxysmal, persistent, longstanding persistent or newly-diagnosed AF prior to admittance for cardiac surgery
* Patients will have elective coronary surgery planned Able of providing informed consent

Exclusion Criteria:

* Patients ≥70 years of age
* Pregnancy Patients with contraindications for oral anticoagulant agents
* Patients undergoing emergency operation
* Patients undergoing concomitant valve replacement
* Severely enlarged LA (>50 mm) on echocardiography
* Prior AF ablation or AF surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation | one year
  The percentage of patients without a recurrence of AF, without antiarrhythmic drugs (AADs), within a follow-up period of at least 12 months after a stabilisation period of 90 days after the initial procedure. An episode of AF is defined as an episode of at least 30 seconds duration.

SECONDARY OUTCOMES:
Duration of hospitalization | One year
  Secondary objectives include the duration of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Marcoen Scholten, MD PhD, Principal Investigator — Medisch Spectrum Twente
Locations (1):
- Medisch Spectrum Twente, Enschede, Overijssel, Netherlands